CLINICAL TRIAL: NCT02735135
Title: Comparison of 2 Mattresses for the Prevention of Bedsores, AIRSOFT DUO and SENTRY 1200 A PRESSION CONSTANTE, by Measuring Skin Pressure in the Sacral Area - a Multicenter Crossover Study
Brief Title: Comparison of 2 Mattresses for the Prevention of Bedsores by Measuring Skin Pressure in the Sacral Area
Acronym: SPA2-ARSFT-DUO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: methodological difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Annie Bauer Confort (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2016/CEDMH-01; 2016-A00188-43 (Other: RCB number)
Record Dates: First submitted 2016-04-07; First posted 2016-04-12 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Pressure Ulcer
Keywords: bedridden
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Airsoft Duo First (Experimental): Patients randomized to this arm will be placed on an AIRSOFT DUO mattress for day 0. They will then be switched to a SENTRY 1200 mattress until the end of month 1.
  Intervention: AIRSOFT DUO for 1 day Intervention: SENTRY 1200 for 1 month
  Interventions: Device: AIRSOFT DUO for 1 day; Device: SENTRY 1200 for 1 month
- SENTRY 1200 First (Experimental): Patients randomized to this arm will be placed on a SENTRY 1200 mattress for day 0. They will then be switched to an AIRSOFT DUO mattress until the end of month 1.
  Intervention: SENTRY 1200 for 1 day Intervention: AIRSOFT DUO for 1 month
  Interventions: Device: SENTRY 1200 for 1 day; Device: AIRSOFT DUO for 1 month

INTERVENTIONS:
Device: AIRSOFT DUO for 1 day — The patient is placed on an AIRSOFT DUO mattress for 1 day.
  Arms: Airsoft Duo First
Device: SENTRY 1200 for 1 month — The patient is placed on a SENTRY 1200 mattress for 1 month.
  Arms: Airsoft Duo First
Device: SENTRY 1200 for 1 day — The patient is placed on a SENTRY 1200 mattress for 1 day.
  Arms: SENTRY 1200 First
Device: AIRSOFT DUO for 1 month — The patient is placed on an AIRSOFT DUO mattress for 1 month.
  Arms: SENTRY 1200 First

SUMMARY:
The main objective of this study is to compare the AIRSOFT DUO and the SENTRY 1200 constant pressure mattresses in terms of peak skin pressures measured at the sacral area.

DETAILED DESCRIPTION:
The secondary objectives of the study are to compare the two devices in terms of:

A. body contact surface area. B. peak pressure at the heel area (combining right and left heels) C. occurrence of pressure ulcers anywhere on the body for 1 month D. patient comfort rated at 1 month (visual analog scale varying from 0-10) E. noise (Likert Scale). F. sleep quality (visual analog scale varying from 0-10).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient spends more than 12 hours in bed and verticalisation is possible
* The patient has a stable medical condition (no complication in the last 10 days) and no visible pressure ulcers
* The patient is at risk for pressure ulcers as assessed by a score ≤ 15 on the Braden Scale
* The patient weighs less than 120 kg

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The subject has a contra-indication for a strictly supine position
* The patient has a knee flexion deformity > 10 °
* The patient is in a state of agitation or refuses to cooperate
* The patient's weight is greater than 120 Kg
* The length of stay is less than one month

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Peak interface pressures at the sacral area (mmHg) | Day 0
Peak interface pressures at the sacral area (mmHg) | Day 1

SECONDARY OUTCOMES:
Body contact surface area (cm^2) | Day 0
Body contact surface area (cm^2) | Day 1
Peak pressure at the heel area (mmHg) | Day 0
Peak pressure at the heel area (mmHg) | Day 1
Pressure ulcer development (yes/no) | Month 1
Self-assessment of comfort by the patient (visual analog scale) | Month 1
Self-assessment for noise (Likert scale) | Month 1
Self-assessment of sleep quality (visual analog scale) | Month 1

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Viollet, MD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - CH de Beziers, Béziers
  - Clinique de Soins de suite et réadaptation Saint Basile, Mougins
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes